CLINICAL TRIAL: NCT00198627
Title: Etiology, Prevention, and Treatment of Neonatal Infections in the Community
Brief Title: Etiology, Prevention and Treatment of Neonatal Infections in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H.22.01.09.05.A1
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Bacterial Infection; Infectious Disease
Keywords: Neonatal bacterial infection
MeSH Terms: conditions — Bacterial Infections; Communicable Diseases | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Co-Trimoxazole; TMP-SMZ

SUMMARY:
The purpose of this study is to determine what are the major types of bacteria that cause newborn infections in the community in rural Bangladesh and whether providing an obstetric and neonatal care package will reduce neonatal deaths by 40%.

DETAILED DESCRIPTION:
The study seeks answers to two questions:

1. What are the major bacterial pathogens responsible for serious neonatal infections in the community in rural Bangladesh?
2. Can provision of a package of obstetric and neonatal care, including active surveillance for serious neonatal illness and referral to hospital, and identification of barriers to care-seeking and design of strategies to address them reduce neonatal mortality rates by at least 40% compared to communities in which such services are not provided?

Despite significant decline in infant and child mortality rates in recent decades, neonatal mortality rates remain unacceptably high. Of the 8 million infant deaths that occur worldwide each year, approximately 4 million occur in the neonatal period.

Hence, the specific aims of the study include:

1. identifying the principal agents of serious bacterial infections in Bangladeshi neonates in the community
2. evaluating the impact of introducing a package of essential obstetric and neonatal care practices in the community, including identifying barriers to care-seeking and design of strategies to address those barriers and
3. building capacity within Bangladesh by training Bangladeshi scientists in epidemiological and microbiological techniques, clinical research methods and best clinical practice through an on-going collaboration with Dhaka Shishu (Children) Hospital and the International Centre for Diarrhoeal Disease Research, Bangladesh.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women (any age)
* newborns

Exclusion Criteria:

* children (outside newborn period)

Min Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16359
Dates: Start 2003-12; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Health workers will visit households at three month intervals for 18 months and survey the status of the babies.

SECONDARY OUTCOMES:
At anytime during the study, if the baby shows symptoms of serious infection, the health worker will offer advice on where to go for treatment, or offer to treat the baby at home.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Darmstadt, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Dhaka Shishu Hospital, Dhaka, Bangladesh

REFERENCES:
- [Derived] Darmstadt GL, Baqui AH, Choi Y, Bari S, Rahman SM, Mannan I, Ahmed AS, Saha SK, Seraji HR, Rahman R, Winch PJ, Chang S, Begum N, Black RE, Santosham M, Arifeen SE; Bangladesh Projahnmo-2 (Mirzapur) Study. Validation of a clinical algorithm to identify neonates with severe illness during routine household visits in rural Bangladesh. Arch Dis Child. 2011 Dec;96(12):1140-6. doi: 10.1136/archdischild-2011-300591. Epub 2011 Sep 30. PMID 21965811
- [Derived] Darmstadt GL, Choi Y, Arifeen SE, Bari S, Rahman SM, Mannan I, Seraji HR, Winch PJ, Saha SK, Ahmed AS, Ahmed S, Begum N, Lee AC, Black RE, Santosham M, Crook D, Baqui AH; Bangladesh Projahnmo-2 Mirzapur Study Group. Evaluation of a cluster-randomized controlled trial of a package of community-based maternal and newborn interventions in Mirzapur, Bangladesh. PLoS One. 2010 Mar 24;5(3):e9696. doi: 10.1371/journal.pone.0009696. PMID 20352087
- [Derived] Darmstadt GL, Saha SK, Choi Y, El Arifeen S, Ahmed NU, Bari S, Rahman SM, Mannan I, Crook D, Fatima K, Winch PJ, Seraji HR, Begum N, Rahman R, Islam M, Rahman A, Black RE, Santosham M, Sacks E, Baqui AH; Bangladesh Projahnmo-2 (Mirzapur) Study Group. Population-based incidence and etiology of community-acquired neonatal bacteremia in Mirzapur, Bangladesh: an observational study. J Infect Dis. 2009 Sep 15;200(6):906-15. doi: 10.1086/605473. PMID 19671016